CLINICAL TRIAL: NCT03179982
Title: Integrated Prevention of HIV Risk and Intimate Partner Violence Among Adolescents in South Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Medical Research Council, South Africa (Other); Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Caroline Kuo, Assistant Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R34MH113484 (NIH)
Record Dates: First submitted 2017-06-01; First posted 2017-06-07 (Actual); Results first posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Sexual Behavior; Intimate Partner Violence
MeSH Terms: conditions — Sexual Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Male adolescents (15-17 years) will be randomly allocated to an intervention arm based on permuted blocked randomization. The intervention arm will receive the HIV-IPV intervention called Safe South Africa.
  Safe South Africa is a group-based, facilitated behavioral intervention for prevention of HIV risk and IPV perpetration specifically tailored for male adolescents. The behavioral intervention is comprised of 2-hour sessions, held once a week for a total of two weeks.
  Interventions: Behavioral: Safe South Africa
- Control (No Intervention): Male adolescents (15-17 years) will be randomly allocated to a control arm based on permuted blocked randomization. The control arm will consist of ordinary usual care. The ordinary usual care condition will consist of a packet of existing available brochures on HIV and other sexually transmitted diseases including testing, prevention, and treatment; IPV prevention and intervention; and places to access prevention, care, and support for these outcomes and related health outcomes.

INTERVENTIONS:
Behavioral: Safe South Africa — Core components of the Safe South Africa intervention include the following:
  * Theory driven, best-evidence intervention approaches to adolescent HIV prevention
  * Linkages between HIV and IPV
  * Victim Empathy
  * Healthy Norms Regarding Masculinity
  * Bystander Intervention Skills
  Arms: Intervention

SUMMARY:
The purpose of this study is to test the feasibility and acceptability of Safe South Africa, an integrated intervention for preventing HIV and Intimate Partner Violence perpetration for male adolescents 15-17 years of age.

DETAILED DESCRIPTION:
This study will investigate the acceptability and feasibility of Safe South Africa, an integrated intervention to prevent adolescent behavioral risk for human immunodeficiency virus (HIV) and perpetration of intimate partner violence (IPV). Safe South Africa is a theory-driven, developmentally-tailored and gender-specific intervention designed for male adolescents 15-17 years of age. The research will be conducted in South Africa, a country with the largest HIV epidemic and some of the highest rates of IPV perpetration in the world. Preventive interventions are urgently needed during adolescence when risk for human immunodeficiency virus (HIV) and intimate partner violence (IPV) increases exponentially. Yet, few behavioral interventions integrate HIV-IPV prevention and are tailored for the unique age and developmental needs of adolescents. We will investigate the acceptability and feasibility of Safe South Africa with three study aims: (1) a development aim - this aim will result in the creation of Safe South Africa, an integrated male adolescent preventive intervention for HIV risk behavior and IPV perpetration; (2) an acceptability aim - this aim will consist of an evaluation of the social ecology of HIV and IPV risk with a survey of N=100 of adolescents, and a test of the acceptability of Safe South Africa through an open pilot trial with N=20 male adolescents; and (3) a feasibility aim - this aim will consist of a randomized controlled pilot trial with 1- and 6-month follow-up in a sample of N=60 male adolescents to assess the feasibility and acceptability for a future fully powered randomized controlled trial to evaluate efficacy of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Male adolescent
* 15-17 years of age, inclusive of 15 and 17

Exclusion Criteria:

* parent/guardian does not provide consent
* adolescent does not provide assent

Ages: 15 Years to 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Participants must identify as male
Enrollment: 60 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-10-23 (Actual); Study Completion 2021-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- South African Medical Research School, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Male adolescents (15-17 years) will be randomly allocated to an intervention arm based on permuted blocked randomization. The intervention arm will receive the HIV-IPV intervention called Safe South Africa.
  Safe South Africa is a group-based, facilitated behavioral intervention for prevention of HIV risk and IPV perpetration specifically tailored for male adolescents. The behavioral intervention is comprised of 2-hour sessions, held once a week for a total of two weeks.
  Safe South Africa: Core components of the Safe South Africa intervention include the following:
  * Theory driven, best-evidence intervention approaches to adolescent HIV prevention
  * Linkages between HIV and IPV
  * Victim Empathy
  * Healthy Norms Regarding Masculinity
  * Bystander Intervention Skills
Period: Overall Study
Arm/Group | Intervention | Control
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30 | 30 | 60
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] — Age in years as reported by participants
  years | 16 [15 to 17] | 16 [15 to 17] | 16 [15 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 30 | 30 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 30 | 30 | 60
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Africa | 30 | 30 | 60
Intimate Partner Violence (IPV) Behavior [Count of Participants; unit: Participants] — Perpetration of sexual violence was assessed using Mary Koss's Sexual Experiences Survey - Short Form Perpetration (SES-SFP).
  This 10-item measure captures frequency of attempted or completed sexual acts for vaginal sex and other forms of sexual contact, methods for perpetration, and if participants view these acts as rape.
  The measure allows for you to calculate the percentage of the sample who has completed 1 or more acts of forced sex (for example, 40% of the sample has engaged in 1 or more acts of forced sex). This is the type of analysis presented in the study.
  Participants | 7 | 6 | 13
Sexual risk behavior - refusal of sex [Count of Participants; unit: Participants] — This is a self reported behavior - refusal of sex - relating to risk for acquisition of HIV
  Participants | 17 | 17 | 34
Likelhood of Bystander Intervention Behavior [Mean (Full Range); unit: score on a scale] — The likelihood of engaging as an active bystander to stop violence is measured through the Bystander Behavior Scale, ranging from 1-40. The questions are answered on a 5-point Likert scale, ranging from 5 = "Very unlikely" to 1 = "Very likely". Lower scores correspond to more likelihood of intervening as an active bystander to stop violence, a measure developed by Miller E, Tancredi DJ, McCauley HL, Decker MR, Virata MCD, Anderson HA, et al. "Coaching Boys into Men": A Cluster-Randomized Controlled Trial of a Dating Violence Prevention Program. Journal of Adolescent Health. 2012;51(5):431-8.
  score on a scale | 29 [25 to 33] | 31 [28 to 35] | 30 [25 to 35]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Satisfaction With Intervention Content
Description: Satisfaction with intervention content is based off of a measure called the Client Satisfaction Questionnaire developed by Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: Development of a general scale. Evaluation and Program Planning. 1979;2:197-207.
  We focus on the question from that scale that assesses satisfaction with the program. The item asks, "How satisfied are you with the program you have received?" Participants could rank their satisfaction from: 1 = quite dissatisfied, 2 = mildly dissatisfied, 3 = mostly satisfied, 4 = very satisfied." Higher scores correspond with higher satisfaction with the intervention program.
Time Frame: 6 months
Population: Those exposed to the intervention were asked about acceptability.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 30
Participants | 28

2. Primary Outcome: Intervention Feasibility
Description: Feasibility is measured by ability to recruit the planned number of participants into the trial. We wanted to recruit at least 95% of the target number of planned participants.
  Feasibility is also measured by retention of trial participants at the final timepoint. A cut off of 75% retention of all participants enrolled in the trial at the final timepoint is viewed as a good result for feasibility.
Time Frame: 6 months
Population: We looked at retention over the trial timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 30 | 30
Participants | 30 | 30

3. Primary Outcome: Intervention Fidelity
Description: Fidelity was not based off a published measure. Rather, a neutral observer rated the facilitator's delivery skills and adherence to a manualized protocol for delivering the intervention that guided the consistent delivery of core theoretical components of the intervention. This neutral observer used the following rankings on a scale with rankings ranging from 1 (equating to a category labeled as low demonstration of skills, <25% of the time) to 3 (equating to a category labeled as high demonstration of skills, >75% of the time). An average ranking of 2.5 or more is seen as success for fidelity.
Time Frame: From the start of the intervention delivery period to the end of the delivery period - a 2 month timespan in total.
Population: We coded interventionist fidelity for core components of delivery to the intervention for those participating in the intervention using rankings on a scale ranging from 1 to 3
Measure: Mean (Full Range); unit: rankings on a scale ranging from 1 to 3
Arm/Group | Intervention
Number analyzed (Participants) | 30
rankings on a scale ranging from 1 to 3 | 2.75 [1 to 3]

4. Secondary Outcome: Number of Participants Who Refused Sex at 6 Months
Description: Measured by comparing whether % of those who refused sex at 6 months versus baseline.
Time Frame: 6 months
Population: This study was not powered to determine efficacy but to look at promising direction of behavior change, and to generate data to inform effect sizes for a future fully powered efficacy trial.
Measure: Count of Participants; unit: Participants
Groups:
- Control: Control participants received a control of nothing.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 30 | 30
Participants | 24 | 24

5. Secondary Outcome: Number of Participants Engaging in Intimate Partner Violence at 6 Months
Description: Measured by examining whether the prevalence of those engaging in intimate partner violence (forced vaginal sex) was significantly lower at 6 months as compared to baseline.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Control Arm: Participants allocated to the control arm received a control of nothing.
Arm/Group | Intervention | Control Arm
Number analyzed (Participants) | 30 | 30
Participants | 0 | 4

6. Secondary Outcome: Change From Baseline in Likelihood of Bystander Intervention Behavior
Description: The likelihood of engaging as an active bystander to stop violence is measured through the Bystander Behavior Scale, ranging from 1-40. The questions are answered on a 5-point Likert scale, ranging from 5 = "Very unlikely" to 1 = "Very likely". Lower scores correspond to more likelihood of intervening as an active bystander to stop violence, a measure developed by Miller E, Tancredi DJ, McCauley HL, Decker MR, Virata MCD, Anderson HA, et al. "Coaching Boys into Men": A Cluster-Randomized Controlled Trial of a Dating Violence Prevention Program. Journal of Adolescent Health. 2012;51(5):431-8.
Time Frame: 6 months
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 30 | 30
score on a scale | 27 [1 to 40] | 30 [1 to 40]

ADVERSE EVENTS:
Time Frame: 6 months
Description: We monitored any serious adverse event and adverse events including injury, death, and other harms.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-04-25): https://cdn.clinicaltrials.gov/large-docs/82/NCT03179982/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-13): https://cdn.clinicaltrials.gov/large-docs/82/NCT03179982/ICF_001.pdf